CLINICAL TRIAL: NCT05041985
Title: Clinical Efficacy of Diazepam After Whiplash
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edin Mešanović (Other)
Responsible Party: Sponsor-Investigator, Edin Mešanović, orthopedic surgeon, Cantonal Hospital Dr. Safet Mujic Mostar
Organization: Cantonal Hospital Dr. Safet Mujic Mostar (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1703016
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2021-09

CONDITIONS: Whiplash Injuries; Whiplash Injury of Cervical Spine
Keywords: whiplash; cervical spine; neck; whiplash injury; muscle spasm; diazepam; muscle strain
MeSH Terms: conditions — Whiplash Injuries; Spasm; Sprains and Strains | interventions — Diazepam

STUDY DESIGN:
Intervention Model Description: Study group will get the recommendation to use one Diazepam 5 mg pill per day (bedtime) for 7 days after whiplash injury.
Who Masked: Investigator
Masking Description: Patients were presented with a sealed opaque envelope which contained a piece of A4 paper with inscriptions Group A or Group B. After choosing one envelope they would tell the nurse which letter they got without the assessor's knowing the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (the Test group) (Experimental): arm which received Diazepam 5 mg therapy for 7 days after whiplash
  Interventions: Drug: Diazepam Tablets
- group B (the control group) (No Intervention): a group which did not receive Diazepam 5 mg therapy

INTERVENTIONS:
Drug: Diazepam Tablets — Diazepam 5 mg tablet once per day (bedtime) for 7 days
  Arms: group A (the Test group)

SUMMARY:
Whiplash injury is very common and lot of patients which suffered the injury have chronic symptoms despite different treatment options. One of main symptoms include muscle spasm and pain caused by neck movement. Diazepam is a well known drug which can be used to treat muscle spasms. The aim of this study is to determine whether short term Diazepam therapy can have positive effect on long term outcomes after whiplash injury.

DETAILED DESCRIPTION:
This randomized, assessor-blinded study was conducted on patients presented due to a cervical spine injury caused by a traffic accident in the previous 48 hours from 1st January 2020 to 31st December 2020. All the patient which were included in this study were divided into 2 groups: group A, the Test group, and group B, the control group. All patients signed the consent to participate in the study prior to randomization. During the initial examination a detailed history was taken and it included Visual Analog Pain Scale (VAS). On follow up examinations 7 days, 6 weeks and 6 months after the injury, all patients completed Neck disability index (NDI), Whiplash disability questionnaire (WDQ) as well as Visual Analog Pain Scale (VAS). Any patient which didn't complete all the follow up examination was excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffered cervical spine injury caused by a traffic accident in the previous 48 hours

Exclusion Criteria:

* younger than 18 years of age; older than 70 years of age; the presence of associated injuries; previous surgery on the cervical spine; previously diagnosed arthrosis of the cervical spine; the presence of a malignant process and previous cervical spine injuries; history of Diazepam allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change in Whiplash Disability Questionnaire score 6 months after injury (0-130; 0 no disability, 130 maximal disability) | 6 months
  Comparation of same score at the follow up examination 7 days after the injury
change in Neck Disability Index score 6 months after injury (0-50, 0 - no disability 50 maximal disability) | 6 months
  Comparation of same score at the follow up examination 7 days after the injury

SECONDARY OUTCOMES:
changes in Visual Analog Scale scores 7 days after the injury (0-10; 0-no pain 10 maximum pain level) | 7 days
  Comparation of same score at the initial examination after the injury
changes in Visual Analog Scale scores 6 weeks after the injury (0-10; 0-no pain 10 maximum pain level) | 6 weeks
  Comparation of same score at the initial examination after the injury
changes in Visual Analog Scale scores 6 months after the injury (0-10; 0-no pain 10 maximum pain level) | 6 months
  Comparation of same score at the initial examination after the injury
change in Whiplash Disability Questionnaire score 6 weeks after injury (0-130; 0 no disability, 130 maximal disability) | 6 weeks
  Comparation of same score at the follow up examination 7 days after the injury
change in Neck Disability Index score 6 weeks after injury (0-50, 0 - no disability 50 maximal disability) | 6 weeks
  Comparation of same score at the follow up examination 7 days after the injury

CONTACTS AND LOCATIONS:
Locations (1):
- KB "dr.Safet Mujic", Mostar, HNK, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
I am ready to share all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: I would be ready to share the IPD after publication.
Access Criteria: I would like to be included in process of who is getting the IPD.

REFERENCES:
- [Background] Spitzer WO, Skovron ML, Salmi LR, Cassidy JD, Duranceau J, Suissa S, Zeiss E. Scientific monograph of the Quebec Task Force on Whiplash-Associated Disorders: redefining "whiplash" and its management. Spine (Phila Pa 1976). 1995 Apr 15;20(8 Suppl):1S-73S. No abstract available. PMID 7604354
- [Background] Uehara Benites MA, Perez-Garrigues H, Morera Perez C. [Clinical symptoms of equilibrium disorders in patients with whiplash syndrome]. Acta Otorrinolaringol Esp. 2009 May-Jun;60(3):155-9. Spanish. PMID 19558900
- [Background] Tanaka N, Atesok K, Nakanishi K, Kamei N, Nakamae T, Kotaka S, Adachi N. Pathology and Treatment of Traumatic Cervical Spine Syndrome: Whiplash Injury. Adv Orthop. 2018 Feb 28;2018:4765050. doi: 10.1155/2018/4765050. eCollection 2018. PMID 29682354
- [Background] Benoist M, Rouaud JP. Whiplash: myth or reality? Joint Bone Spine. 2002 Jun;69(4):358-62. doi: 10.1016/s1297-319x(02)00410-4. No abstract available. PMID 12184430